CLINICAL TRIAL: NCT07193641
Title: A Prospective, Single-Arm Phase II Clinical Trial of Standard Systemic Therapy Combined With Spatial Fractionated Radiotherapy (SFRT) for Oligoprogressive Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study on Using SFRT With Standard Treatment for Oligoprogressive NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y202-0552
Record Dates: First submitted 2025-08-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: oligoprogressive NSCLC; SFRT; systemic therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SFRT plus systemic therapy (Experimental)
  Interventions: Radiation: Spatially Fractionated Radiotherapy (SFRT)+Stereotactic Body Radiation Therapy (SBRT); Drug: The systemic therapy

INTERVENTIONS:
Radiation: Spatially Fractionated Radiotherapy (SFRT)+Stereotactic Body Radiation Therapy (SBRT) — The intervention includes SFRT for larger oligoprogressive lesions (≥4.5 cm in diameter), utilizing image-guided CT, including 4D-CT, with Lattice technique planning. The dose fractionation will be determined by the radiation oncologist based on clinical parameters, with peak doses ranging from 6-15 Gy/Fx and valley doses from 1.8-4 Gy/Fx, typically in 1-5 fractions.
  For smaller oligoprogressive lesions, stereotactic body radiotherapy (SBRT) or intensity-modulated radiotherapy (IMRT) will be selected based on clinical parameters.
Drug: The systemic therapy — Continuation or switch of prior standard regimen (chemotherapy, targeted TKI, or PD-1/PD-L1 inhibitor) at investigator discretion until further progression or intolerable toxicity.

SUMMARY:
The goal of this clinical trial is to learn if spatially fractionated radiotherapy (SFRT) combined with standard systemic therapy can treat oligoprogressive non-small cell lung cancer (NSCLC) in patients who have progressed after at least one line of systemic therapy. The main question it aims to answer is:

- Can the combination of SFRT and standard systemic therapy improve progression-free survival (PFS) compared to standard systemic therapy alone?

Participants will:

* Undergo SFRT treatment for oligoprogressive lesions, with specific dose fractionation determined by the radiation oncologist based on clinical parameters.
* Continue their standard systemic therapy, which may include chemotherapy, targeted therapy, or immunotherapy, as adjusted by their treating physician.
* Have regular follow-up assessments, including imaging studies to evaluate treatment response and monitor for disease progression.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older, regardless of sex.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less, with an expected survival of more than 3 months.
* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) with oligometastatic disease (up to 5 separate progressive lesions), having received and progressed after at least one line of systemic therapy (chemotherapy, targeted therapy, or immunotherapy).
* The target lesion for radiotherapy has not been previously irradiated, or it has been more than 6 months since the last radiotherapy.
* The diameter of the target lesion is at least 4.5 cm, suitable for lattice radiotherapy planning.
* No new or enlarged brain metastases; if brain metastases were previously treated with standard radiotherapy, they must be stable.
* Adequate hematologic and biochemical profiles, including hemoglobin ≥9.0 g/dL, absolute neutrophil count (ANC) ≥1500/mm³, platelet count ≥100,000/mm³, total bilirubin ≤1.5 times the upper limit of normal (ULN) (or direct bilirubin ≤ULN if total bilirubin >1.5 times ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times ULN (or ≤5 times ULN if liver involvement is present), and creatinine ≤1.5 times ULN (or glomerular filtration rate [GFR] >60 mL/min if creatinine >1.5 times ULN).
* For women of childbearing potential, a negative pregnancy test within 7 days prior to registration.

Exclusion Criteria

* Presence of other systemic diseases or severe comorbidities that the investigator believes would make the patient unsuitable for the study or significantly interfere with the assessment of the safety and toxicity of the study regimen.
* Active autoimmune diseases requiring systemic treatment, or a history of severe autoimmune diseases, such as interstitial lung disease.
* Uncontrolled concurrent diseases, including but not limited to: infections requiring systemic treatment, active tuberculosis (TB), severe or chronic gastrointestinal diseases associated with diarrhea (e.g., Crohn's disease), active hepatitis B (defined by positive hepatitis B surface antigen [HBsAg]), active hepatitis C (defined by positive hepatitis C virus [HCV] RNA), symptomatic congestive heart failure, unstable angina, unstable cardiac arrhythmias, myocardial infarction within the past 6 months, or congestive heart failure requiring continuous maintenance therapy for life-threatening ventricular arrhythmias.
* Mental illness or social situations that might limit the patient's ability to comply with study requirements (e.g., drug abuse).
* Participation in other interventional clinical trials with experimental drugs that could be considered treatment for the primary tumor.
* Allergy to immunotherapy drugs, or discontinuation of immunotherapy drugs due to adverse events in the past, or grade 3 or higher immune-related adverse events during previous immunotherapy, or any grade of immune-related neurological or ocular adverse events.
* History of other active malignancies within the past 6 months, except for non-melanoma skin cancer, papillary thyroid cancer, prostate cancer, or cervical carcinoma in situ that have been treated with curative intent and are currently considered to have a recurrence risk of less than 30%.
* History of allogeneic organ transplantation or active primary immunodeficiency.
* Any other condition that the investigator deems a valid reason for exclusion, such as potential situations inconsistent with the clinical protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From date of first study treatment to documented progression or death, assessed at 6 weeks, 12 weeks, 24 weeks, 48 weeks, and 72 weeks.
  PFS will be determined based on radiological assessments using CT or MRI scans, according to the RECIST v1.1 criteria. Disease progression will be defined as an increase of at least 20% in the size of target lesions or the appearance of new lesions.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) of Irradiated Lesions | 1 month after the completion of SFRT treatment and then every 3 months thereafter
  ORR will be assessed using RECIST v1.1 criteria. ORR includes complete response (CR) and partial response (PR). Tumor response will be evaluated through radiological imaging (CT or MRI) of the irradiated lesions
Treatment-Related Adverse Events (TRAEs) | throughout the treatment period and for a predefined follow-up period, typically up to 12 months after treatment completion
  TRAEs will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The incidence and severity of adverse events will be recorded at each follow-up visit, with a focus on grade 3 or higher events
Overall Survival (OS) | From date of first study treatment to death from any cause, assessed at 24 weeks, 48 weeks, and 72 weeks.
  OS will be determined based on the date of death recorded in medical records or through follow-up contacts with patients or their families

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Hangzhou, Zhejiang, China